CLINICAL TRIAL: NCT05075590
Title: Coronary ANgiography and ACCESS Following Implantation of a Supra-Annular Transcatheter Heart Valve With Commissural Alignment: The CAN-ACCESS Pilot Study
Brief Title: Coronary Access After Supra-Annular THV Implantation
Acronym: CAN-ACCESS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Medtronic (Industry); The Centre for Cardiovascular Innovation - Centre d'Innovation Cardiovasculaire (CCI-CIC) (Unknown)
Responsible Party: Principal Investigator, David Wood, Interventional and Structural Cardiologist, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H21-01704
Record Dates: First submitted 2021-09-14; First posted 2021-10-13 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Coronary Angiography; Transcatheter Aortic Valve Replacement
Keywords: elective transfemoral TAVR; Evolut valve; Supra-Annular Transcatheter Heart Valve; Commissural Alignment; Coronary Angiography; Transcatheter Aortic Valve Replacement; Coronary Access
MeSH Terms: interventions — Coronary Angiography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Diagnostic Test: Coronary Angiography — Following TAVR, the operators will attempt to selectively engage both the right and left coronary arteries. Catheter choice and engagement technique will be at the discretion of the operator.

SUMMARY:
To determine the optimal technique and equipment for selective coronary engagement specifically following Evolut THV implantation using commissural alignment.

DETAILED DESCRIPTION:
Patients will undergo elective transfemoral TAVR with the Evolut THV. The operators will attempt to selectively engage both the right and left coronary arteries through standardized angiographic views. The CCI-CIC CoreLabs will adjudicate angiographic views, post-TAVR CT scan, and determine if the coronaries were selectively engaged. Catheter choice, adjunctive tools if needed (e.g guide extension, wires etc) and engagement technique will be at the discretion of the operator. All images and fluoroscopic views will be anonymized, saved and imported to the CCI-CIC Angiographic and CT CoreLabs.

Statistical analysis:

Patient baseline and outcome data will be presented as mean and standard deviation (SD) for normally distributed variables, median and interquartile range (IQR) for non-normally distributed variables, and frequency and proportion for categorical variables.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing elective transfemoral TAVR with the Evolut THV (Medtronic, Minneapolis, MN, USA).
2. Written informed consent to participate in the study.

Exclusion Criteria:

1. Hemodynamic or respiratory instability immediately prior to TAVR or during TAVR.
2. Advanced chronic kidney disease, defined as a GFR <30 ml/min.
3. Valve-in-valve TAVR
4. Prior CABG
5. Aorto-ostial coronary artery disease.
6. Prior PCI of the left main or right coronary ostium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-10-27 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
The ability to selectively engage and obtain diagnostic epicardial coronary angiography images from the right and left coronary ostia | Immediately post-TAVR
  Coronary engagement will be classified as:
  1. Partially successful if non-selective engagement is achieved (catheter is unable to be placed in the coronary ostia) and there is adequate opacification of the coronary vessels.
  2. Successful if selective engagement is achieved with placement of the coronary catheter in the coronary ostia and adequate opacification of the coronary vessels.
  3. Unsuccessful if engagement is not possible and there is insufficient opacification of the coronary vessels.

SECONDARY OUTCOMES:
Total fluoroscopic time (mins) from catheter insertion to selective coronary engagement. | During TAVR procedure
Total contrast use (ml) from catheter insertion to selective coronary engagement. | During TAVR procedure
Type of wire and catheter used for successful right and left coronary engagement | During TAVR procedure
  Reporting of the wire and catheter type will be collected
Total number and types of wires and catheters used. | During TAVR procedure
Description of type of technique utilized to achieve selective coronary engagement. | During TAVR procedure
  Report of description will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Janarthanan Sathananthan, MBChB, MPH, Principal Investigator — University of British Columbia
Locations (4):
- UPMC Harrisburg, Harrisburg, Pennsylvania, United States
- Canada (3):
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

REFERENCES:
- [Result] Pilgrim T, Windecker S. Expansion of transcatheter aortic valve implantation: new indications and socio-economic considerations. Eur Heart J. 2018 Jul 21;39(28):2643-2645. doi: 10.1093/eurheartj/ehy228. No abstract available. PMID 29701845
- [Result] Mack MJ, Leon MB, Thourani VH, Makkar R, Kodali SK, Russo M, Kapadia SR, Malaisrie SC, Cohen DJ, Pibarot P, Leipsic J, Hahn RT, Blanke P, Williams MR, McCabe JM, Brown DL, Babaliaros V, Goldman S, Szeto WY, Genereux P, Pershad A, Pocock SJ, Alu MC, Webb JG, Smith CR; PARTNER 3 Investigators. Transcatheter Aortic-Valve Replacement with a Balloon-Expandable Valve in Low-Risk Patients. N Engl J Med. 2019 May 2;380(18):1695-1705. doi: 10.1056/NEJMoa1814052. Epub 2019 Mar 16. PMID 30883058
- [Result] Asgar AW, Ouzounian M, Adams C, Afilalo J, Fremes S, Lauck S, Leipsic J, Piazza N, Rodes-Cabau J, Welsh R, Wijeysundera HC, Webb JG. 2019 Canadian Cardiovascular Society Position Statement for Transcatheter Aortic Valve Implantation. Can J Cardiol. 2019 Nov;35(11):1437-1448. doi: 10.1016/j.cjca.2019.08.011. PMID 31679616
- [Result] Nishimura RA, Otto CM, Bonow RO, Carabello BA, Erwin JP 3rd, Fleisher LA, Jneid H, Mack MJ, McLeod CJ, O'Gara PT, Rigolin VH, Sundt TM 3rd, Thompson A. 2017 AHA/ACC Focused Update of the 2014 AHA/ACC Guideline for the Management of Patients With Valvular Heart Disease: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. J Am Coll Cardiol. 2017 Jul 11;70(2):252-289. doi: 10.1016/j.jacc.2017.03.011. Epub 2017 Mar 15. No abstract available. PMID 28315732
- [Result] Htun WW, Grines C, Schreiber T. Feasibility of coronary angiography and percutaneous coronary intervention after transcatheter aortic valve replacement using a Medtronic self-expandable bioprosthetic valve. Catheter Cardiovasc Interv. 2018 Jun;91(7):1339-1344. doi: 10.1002/ccd.27346. Epub 2017 Oct 8. PMID 28988450
- [Result] Yudi MB, Sharma SK, Tang GHL, Kini A. Coronary Angiography and Percutaneous Coronary Intervention After Transcatheter Aortic Valve Replacement. J Am Coll Cardiol. 2018 Mar 27;71(12):1360-1378. doi: 10.1016/j.jacc.2018.01.057. PMID 29566822
- [Result] Boukantar M, Gallet R, Mouillet G, Belarbi A, Rubimbura V, Ternacle J, Dubois-Rande JL, Teiger E. Coronary Procedures After TAVI With the Self-Expanding Aortic Bioprosthesis Medtronic CoreValve, Not an Easy Matter. J Interv Cardiol. 2017 Feb;30(1):56-62. doi: 10.1111/joic.12363. Epub 2017 Jan 11. PMID 28078734
- [Result] Blumenstein J, Kim WK, Liebetrau C, Gaede L, Kempfert J, Walther T, Hamm C, Mollmann H. Challenges of coronary angiography and intervention in patients previously treated by TAVI. Clin Res Cardiol. 2015 Aug;104(8):632-9. doi: 10.1007/s00392-015-0824-5. Epub 2015 Feb 27. PMID 25720330
- [Result] Barbanti M, Costa G, Picci A, Criscione E, Reddavid C, Valvo R, Todaro D, Deste W, Condorelli A, Scalia M, Licciardello A, Politi G, De Luca G, Strazzieri O, Motta S, Garretto V, Veroux P, Giaquinta A, Giuffrida A, Sgroi C, Leon MB, Webb JG, Tamburino C. Coronary Cannulation After Transcatheter Aortic Valve Replacement: The RE-ACCESS Study. JACC Cardiovasc Interv. 2020 Nov 9;13(21):2542-2555. doi: 10.1016/j.jcin.2020.07.006. Epub 2020 Oct 14. PMID 33069648
- [Result] Abdelghani M, Landt M, Traboulsi H, Becker B, Richardt G. Coronary Access After TAVR With a Self-Expanding Bioprosthesis: Insights From Computed Tomography. JACC Cardiovasc Interv. 2020 Mar 23;13(6):709-722. doi: 10.1016/j.jcin.2020.01.229. PMID 32192691
- [Result] Tang GHL, Zaid S, Fuchs A, Yamabe T, Yazdchi F, Gupta E, Ahmad H, Kofoed KF, Goldberg JB, Undemir C, Kaple RK, Shah PB, Kaneko T, Lansman SL, Khera S, Kovacic JC, Dangas GD, Lerakis S, Sharma SK, Kini A, Adams DH, Khalique OK, Hahn RT, Sondergaard L, George I, Kodali SK, De Backer O, Leon MB, Bapat VN. Alignment of Transcatheter Aortic-Valve Neo-Commissures (ALIGN TAVR): Impact on Final Valve Orientation and Coronary Artery Overlap. JACC Cardiovasc Interv. 2020 May 11;13(9):1030-1042. doi: 10.1016/j.jcin.2020.02.005. Epub 2020 Mar 16. PMID 32192985